CLINICAL TRIAL: NCT05280223
Title: Dexmedetomidine Versus Hyalase Local Injection for Pain Alleviation in Patients With Carpal Tunnel Syndrome; A Randomized Clinical Trial
Brief Title: Dexmedetomidine Versus Hyalase Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB0002022
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Carpal Tunnel Syndrome; Pain, Chronic
MeSH Terms: conditions — Carpal Tunnel Syndrome; Chronic Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmeditomidine group (Active Comparator): injection of 1 microgram/kg dexmedetomidine + 10 cc saline injection nearby median nerve as hydrodissection
  Interventions: Drug: Dexmedetomidine
- Hyalase (Active Comparator): injection of Hyalase + 10 cc saline injection nearby median nerve as hydro-dissection
  Interventions: Drug: Hyalase

INTERVENTIONS:
Drug: Dexmedetomidine — injection of 1 microgram/kg dexmeditomidine + 10 cc saline injection nearby median nerve as hydrodissection
  Arms: Dexmeditomidine group
Drug: Hyalase — injection of Hyalase + 10 cc saline injection nearby median nerve as hydro-dissection
  Arms: Hyalase

SUMMARY:
Carpal tunnel syndrome (CTS) is a common peripheral entrapment neuropathy, this study aims to investigate if, and to what extent hydro-dissection hyalase and saline versus dexmedetomidine upon the median nerve could offer symptoms and clinical improvement

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common compression syndrome the upper extremities. Its problem has a high prevalence ranged estimated prevalence of 3.8% in the general population, 3 and 7.8% in the working population. It occurs at any age, especially in individuals in their 40s to 60s, and the male: female ratio is reported to be 3:7. A lot of treatment modalities have been tried to improve the condition, starting from local anesthetic injection, steroid, and up to surgical decompression of the nerves.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* complaining of carpal tunnel syndrome of 3 month duration or more
* diagnosed axonal neuropathy using electrodiagnosis , nerve conduction study

Exclusion Criteria:

* • patient refusal infection at the site of intervention

  * local anesthetic allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Pain alleviation | 6 months
  pain alleviation improvement of pain measured by visual analog scale , no pain the scale equal zero , and worst pain the scale equal 10

SECONDARY OUTCOMES:
Median nerve cross sectional area | 6 months
  Changes in ultrasound imaging change of cross sectional area in cubic mellimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No